CLINICAL TRIAL: NCT07357610
Title: An Open-Label Drug Interaction Clinical Study to Evaluate Itraconazole, Rifampin, Midazolam and SIM0270 in Chinese Healthy Adult Participants
Acronym: SIM0270-104
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SIM0270-104
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants
MeSH Terms: interventions — Itraconazole; Rifampin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 : to evaluate the effect of the CYP3A4 inhibitor itraconazole on the pharmacokinetics of SI (Experimental): Cohort 1 is planned to enroll 16-20 healthy adult participants, both male and female
  Interventions: Drug: SIM0270; Drug: itraconazole
- Cohort 2: to evaluate the effect of CYP3A4 inducer rifampin on the pharmacokinetics of SIM0270. (Experimental): Cohort 2 is planned to enroll 16-20 healthy adult participants, both male and female.
  Interventions: Drug: SIM0270; Drug: Rifampin
- Cohort 3: to evaluate the effect of SIM0270 on the pharmacokinetics of the CYP3A4 substrate midazol (Experimental): Cohort 3 is planned to enroll 16-20 healthy adult participants，male only
  Interventions: Drug: SIM0270; Drug: midazolam

INTERVENTIONS:
Drug: SIM0270 — oral
Drug: itraconazole — oral
  Arms: Cohort 1 : to evaluate the effect of the CYP3A4 inhibitor itraconazole on the pharmacokinetics of SI
Drug: Rifampin — oral
  Arms: Cohort 2: to evaluate the effect of CYP3A4 inducer rifampin on the pharmacokinetics of SIM0270.
Drug: midazolam — oral
  Arms: Cohort 3: to evaluate the effect of SIM0270 on the pharmacokinetics of the CYP3A4 substrate midazol

SUMMARY:
This study is an open-label, fixed-sequence, two-period Phase 1 clinical trial in healthy adult Chinese participants with a total of 3 cohorts, 16-20 healthy adult Chinese participants are planned to be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* The participant fully understand the test content, process and possible adverse reactions, voluntarily sign informed consent, have good communication with the researchers, and can complete all the test procedures in accordance with the protocol.
* Cohorts 1 and 2: healthy male and female participants aged ≥ 18 and ≤ 55 years; Cohort 3: healthy male participants aged ≥ 18 and ≤ 55 years.
* Male participants weigh ≥ 50 kg; Female participants weigh ≥ 45 kg; Body mass index ≥ 19 kg/m2 and ≤ 26 kg/m2.
* Cohorts 1 and 2: all female participants of childbearing potential and male participants with partners of women of childbearing potential agree to take recognized effective contraceptive measures during the study period and within 6 months after the last dose of the investigational product, starting from signing the informed consent; Cohort 3: male participants with partners of women of childbearing potential agree to take recognized effective contraceptive measures during the study period and within 6 months after the last dose of the investigational product, starting from signing the informed consent.

Exclusion Criteria:

Past/Ongoing Medical History

* Neurological/psychiatric, respiratory, cardiovascular, gastrointestinal, urinary, hematological and lymphatic, endocrine, skeletal-muscular disorders, especially hepatic and renal insufficiency, or any other disease and condition that may affect the results of the study or the safety of the participants.
* History of dysphagia or any gastrointestinal disorder affecting drug absorption.
* Presence of risk factors for Torsade de Pointes (e.g., history of heart failure, hypokalemia, family history of QT prolongation syndrome), or other clinically significant abnormalities judged by the study doctor (including but not limited to: complete left bundle branch block; right bundle branch block; first-, second-, or third-degree heart block; sick sinus syndrome or previous history of myocardial infarction).
* History of active or latent tuberculosis.
* History of malignancy. Except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin cancer, or stage I uterine cancer (disease-free interval of at least 5 years).
* Any acute or chronic condition that, in the opinion of the investigator, would limit the ability of participants to complete and/or participate in this clinical study.

Surgical history • Those who have undergone major surgery within 6 months prior to screening or are scheduled to undergo surgery during the study and are judged by the investigator to be inappropriate for enrollment.

History of allergy

• Allergic to the study drug or any component of the study drug, with a history of specific allergies (asthma, urticaria, eczema, etc.) or allergic constitution (e.g., those allergic to two or more drugs, food such as milk and pollen).

Medication history

* Use of hormone replacement therapy or selective estrogen mediators within 1 year prior to screening.
* Use or planned use of any drug/product within 4 weeks prior to screening that would alter the process of drug absorption, metabolism, or elimination.
* Use of any prescription drugs/products within 2 weeks prior to screening or over-the-counter medications (including vitamins, minerals, phytotherapies, herbal and botanical preparations) within 1 week prior to screening.

Screening or Baseline Examinations

* Laboratory tests, physical examination, vital signs, 12-lead electrocardiogram, chest anterolateral film, abdominal B-ultrasound results were abnormal and clinically significant as judged by the investigator.
* Screening (mean) or baseline ECG heart rate < 60 beats/min or > 100 beats/min, QTcF interval > 450 ms.
* Women of childbearing potential who have a positive pregnancy test or are pregnant or lactating (see Appendix 1 for definitions of women of non-childbearing potential).
* Positive tests for hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV) antibody, treponema pallidum antibody.
* History of drug abuse or positive drug abuse screening.
* Regular drinkers, i.e., on average, more than 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) within 3 months prior to screening or during the screening period to the first dose; Or alcohol breath test positive.
* Those who smoke more than 5 cigarettes per day within 3 months prior to screening or who cannot quit during the trial.
* Participation in any drug clinical trial as a participant and taking study drug or medical device intervention within 3 months prior to screening.
* Consumption of grapefruit or grapefruit-related citrus (e.g., grapefruit) fruit or juice within 1 week prior to screening, or use of alcoholic or caffeinated food or beverages within 72 h prior to screening.
* Those who have special requirements for diet and cannot comply with the diet provided and corresponding regulations.
* Those who have difficulty in venous blood collection, or have a history of fainting blood and needle sickness, or who cannot tolerate venous indwelling needle blood collection.
* Those who have donated blood or lost more than 200 mL of blood within 3 months prior to screening, or have received blood transfusions or blood products within 2 months.
* Participants have other conditions that are not suitable for participation in the study, or participants may not be able to complete the study for other reasons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of SIM0270 | Day 1-Day 13, Day 16-Day 30
  To determine the effect of itraconazole on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Area under concentration curve from time 0 to the last quantifiable concentration (AUC0-t) of SIM0270 | Day 1-Day 13, Day 16-Day 30
  To determine the effect of itraconazole on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Area under concentration-time curve from time 0 to infinity (AUC0-∞) of SIM0270 | Day 1-Day 13, Day 16-Day 30
  To determine the effect of itraconazole on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Area under concentration-time curve from time 0 to tau (AUC0-tau) of SIM0270 | Day 1-Day 13, Day 16-Day 30
  To determine the effect of itraconazole on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Terminal half-life（t1/2）of SIM0270 | Day 1-Day 13, Day 16-Day 30
  To determine the effect of itraconazole on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Maximum observed concentration (Cmax) of SIM0270 | Day 1-Day 13, Day 20-Day 32
  To determine the effect of rifampicin on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Area under concentration curve from time 0 to the last quantifiable concentration (AUC0-t) of SIM0270 | Day 1-Day 13, Day 20-Day 32
  To determine the effect of rifampicin on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Area under concentration-time curve from time 0 to infinity (AUC0-∞) of SIM0270 | Day 1-Day 13, Day 20-Day 32
  To determine the effect of rifampicin on the PK of a single dose of SIM0270 in Chinese healthy adult participants
Terminal half-life（t1/2）of SIM0270 | Day 1-Day 13, Day 20-Day 32
  To determine the effect of rifampicin on the PK of a single dose of SIM0270 in Chinese healthy adult participants.
Maximum observed concentration (Cmax) of midazolam | Day 1-Day 2, Day 11-Day 13
  To determine the effect of SIM0270 on the PK of a single dose of midazolam in Chinese healthy adult male participants.
Area under concentration curve from time 0 to the last quantifiable concentration (AUC0-t) of Midazolam | Day 1-Day 2, Day 11-Day 13
  To determine the effect of SIM0270 on the PK of a single dose of midazolam in Chinese healthy adult male participants.
Area under concentration-time curve from time 0 to infinity (AUC0-∞) of Midazolam | Day 1-Day 2, Day 11-Day 13
  To determine the effect of SIM0270 on the PK of a single dose of midazolam in Chinese healthy adult male participants.
Terminal half-life（t1/2）of midazolam | Day 1-Day 2, Day 11-Day 13
  To determine the effect of SIM0270 on the PK of a single dose of midazolam in Chinese healthy adult male participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University of Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No